CLINICAL TRIAL: NCT04215146
Title: A Study to Assess Overall Response Rate by Inducing an Inflammatory Phenotype in Metastatic BReast cAnCEr With the Oncolytic Reovirus PeLareorEp in CombinaTion With Anti-PD-L1 Avelumab and Paclitaxel - BRACELET-1 Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Collaborators: PrECOG, LLC. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REO 028; PrE0113 (Other: PrECOG, LLC.)
Record Dates: First submitted 2019-12-24; First posted 2020-01-02 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Metastatic
Keywords: Breast; Breast Cancer; Breast Cancer Metastatic; Locally Advanced Breast Cancer; Pelareorep; Avelumab; Paclitaxel; Reovirus; Oncolytic virus; HR+ breast cancer; HER2- breast cancer; Breast malignancy
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; reolysin; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): Patients receive paclitaxel alone.
  Interventions: Drug: Paclitaxel
- Cohort 2 (Experimental): Patients receive pelareorep + paclitaxel.
  Interventions: Drug: Paclitaxel; Biological: Pelareorep
- Cohort 3 (Experimental): Patients receive pelareorep + paclitaxel + avelumab.
  Interventions: Drug: Paclitaxel; Biological: Pelareorep; Drug: Avelumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80 mg/m^2 1-hour IV infusion on days 1, 8, and 15 of a 28-day cycle.
Biological: Pelareorep — Pelareorep 4.5 x 10^10 TCID50 1-hour IV infusion days 1, 2, 8, 9, and 15, 16 of a 28-day cycle.
  Arms: Cohort 2; Cohort 3
Drug: Avelumab — Avelumab 10 mg/kg (not more than 800 mg) 1-hour IV infusion days 3 and 17 of a 28-day cycle.
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to find out the possible anti-cancer effect of pelareorep in combination with chemotherapy [paclitaxel] and avelumab in treating a type of breast cancer called Hormone Receptor positive (HR+)/Human Epidermal Growth Factor Receptor 2 negative(HER2-) breast cancer, which is either locally advanced or has metastasized (cancer that has spread in your body). The study will investigate if pelareorep in combination with paclitaxel and avelumab is more effective than paclitaxel alone, or pelareorep and paclitaxel. The safety of the combination treatments will also be evaluated.

DETAILED DESCRIPTION:
This is an open-label randomized Phase 2, 3-cohort study to evaluate the safety and efficacy of pelareorep, paclitaxel and avelumab in Hormone Receptor+ (HR+)/Human Epidermal Growth Factor Receptor 2 negative (HER2-) with endocrine-refractory metastatic breast cancer.

Patients will be randomized to one of three treatment cohorts: paclitaxel alone, pelareorep + paclitaxel, or pelareorep + paclitaxel + avelumab. A three patient safety run-in will be conducted in the cohort for pelareorep + paclitaxel + avelumab prior to beginning randomization into all three cohorts.

Patients will give mandatory blood samples and optional tumor biopsies, which will be analyzed for biomarkers to determine the immunological changes within the tumor microenvironment and peripheral blood in patients treated with paclitaxel alone, in combination with pelareorep, and in combination with pelareorep and avelumab.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Must have a histological/cytological diagnosis of breast cancer. Disease must be:

   * Positive for estrogen receptor (ER) and/or progesterone receptor (PgR) as defined by

     ≥ 1% tumor cell nuclei immunoreactive.
   * Negative for HER2 amplification / overexpression as defined per the American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines. However, patients with HER2 equivocal disease for whom HER2 targeted therapy isn't indicated are also eligible for enrollment.
3. ECOG performance status of 0-1
4. Must have unresectable locally advanced or metastatic disease, for which no curative therapy exists and for which systemic chemotherapy is indicated.
5. Measurable disease as defined by RECIST Version 1.1
6. Prior Hormonal Therapy:

   * Patients must have progressed on at least 1 hormone-based therapy with a CDK4/6 inhibitor. Patients who received a CDK4/6 inhibitor in the adjuvant setting and progressed while on or within 6 months of discontinuation of CDK4/6 inhibitor therapy are eligible.
   * Prior mTOR inhibitor therapy is allowed but is not required.
7. Ability to understand and willingness to sign IRB-approved informed consent.
8. Willing to provide blood samples for research
9. Adequate organ function as measured by the following criteria, obtained ≤ 2 weeks prior to registration:

   Hematology:
   * Neutrophils ≥ 1.5 x 10^9/L
   * Platelets ≥ 100 x 10^9/L
   * Lymphocytes ≥ 0.8 x 10^9/L
   * INR < 1.5x ULN (Unless on therapeutic anticoagulation)
   * PTT < 1.5x ULN

   Biochemistry:
   * Serum Creatinine ≤ 1.5x ULN
   * Total Bilirubin ≤ 1.0x ULN (unless due to Gilbert's Disease and direct bilirubin <ULN)
   * ALT and AST ≤ 3x ULN (Note: ≤ 5x ULN if documented liver metastasis)
   * Proteinuria ≤ Grade 2* (using spot testing; if Grade 3 repeat with mid-stream urine; if still Grade 3 then urine collection for 24 hours to confirm Grade 0, 1 or 2) *as per National Cancer Institute Common Terminology Criteria for Adverse (NCI-CTCAE)
10. Women must not be pregnant or breastfeeding since we do not know the effects of the study drugs on the fetus or breastfeeding child. All sexually active females of childbearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have a blood test to rule out pregnancy within 2 weeks prior to registration.
11. Sexually active women of child-bearing potential with a non-sterilized male partner must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation, and for 3 months following last dose of study drugs. Method of contraception must be documented. NOTE: If a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Exclusion Criteria:

1. No major surgery within 21 days prior to beginning study treatment. Major surgery >21 days prior to beginning study treatment is permitted provided that the patient has recovered adequately to receive systemic chemotherapy. NOTE: Placement of a vascular access device is not considered major surgery.
2. Patients who have received radiation treatment within 14 days of beginning study treatment are excluded. Patients who have received palliative radiation ≥ 14 days prior to beginning study treatment may enroll if they have recovered from all local and systemic side effects to ≤ Grade 1 (NCI-CTCAE).
3. No prior chemotherapy in the advanced/metastatic setting is allowed. Patients may have received chemotherapy in the (neo)adjuvant setting. Patients receiving (neo)adjuvant taxanes must have a disease-free interval of at least 12 months.
4. No known active, uncontrolled or symptomatic Central Nervous System (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms,cerebral edema, and/or progressive growth. Patients with CNS metastases treated with radiation therapy (Whole-Brain Radiation Therapy [WBXRT] or Stereotactic Radiotherapy [SRS]) are eligible if, >28 days following completion of XRT, they show stable disease on post-treatment MRI/CT, are off corticosteroids, and are neurologically stable.
5. No known history of other malignancies, except for adequately treated non-melanoma skin cancer or solid tumors curatively treated with no evidence of disease for >3 years.
6. Not on chronic immunosuppressive therapy including, but not exclusively, steroids (≥ 10 mg prednisone a day or equivalent) or monoclonal antibodies, chronic methotrexate or cyclophosphamide, tacrolimus or sirolimus.
7. No known HIV infection. Testing not required in absence of clinical suspicion.
8. No known active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection or undergoing anti-viral treatment. Testing for HBV/HCV is not required in absence of clinical suspicion.
9. No concurrent disease or condition that would interfere with study participation or safety,such as any of the following:

   • Active, clinically significant infection either Grade >2 by CTCAE V5.0 or requiring the use of parenteral anti-microbial agents within 14 days before registration.
10. No active or history of any autoimmune disease (patients with diabetes Type 1, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible) or immunodeficiencies.
11. Patients may not have evidence of uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or higher), unstable angina, or myocardial infarction within the past 6 months prior to registration. NOTE: Patients with asymptomatic rate-controlled atrial fibrillation may participate.
12. Patients may not have other significant diseases (for example, inflammatory bowel disease), which, in the opinion of the Investigator, might impair the patient's tolerance of trial treatment.
13. Patients with a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent are not eligible.
14. Patients who have contraindications to treatment with paclitaxel and/or neuropathy >Grade 2 are not eligible.
15. Patients who have not recovered from clinically significant acute toxicities of previous therapy are not eligible, except treatment-related alopecia or stable sensory neuropathy ≤ Grade 2.
16. No prior therapy with any investigational anti-cancer therapy within 30 days. Prior immunotherapies are prohibited.
17. No prior therapy with checkpoint inhibitors (e.g., anti-PD-1/PD-L1 antibodies), checkpoint agonist agents (e.g., anti-GITR, anti-OX40 antibodies) and/or another active immunotherapy in breast cancer such as cancer vaccines or oncolytic virsus.
18. Patients with any serious medical or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of the treatment according to the protocol, are not eligible.
19. Patients with legal incapacity or limited legal capacity are not eligible.
20. Patients with known alcohol or drug abuse are not eligible.
21. Patients may not participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial, throughout the duration of this study.
22. Patients may not have any vaccine, including against SARS-COV-2 (COVID-19) <14 days prior to Cycle 1 Day 1 nor in the first cycle of study treatment. Inactivated vaccines (including against COVID-19 or seasonal influenza) are permitted after the first cycle of study treatment is complete.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2025-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Park, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU/Massey Cancer Center, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel: Patients receive paclitaxel alone.
  Paclitaxel: Paclitaxel 80 mg/m^2 1-hour IV infusion on days 1, 8, and 15 of a 28-day cycle.
- Pelareorep + Paclitaxel: Patients receive pelareorep + paclitaxel.
  Paclitaxel: Paclitaxel 80 mg/m^2 1-hour IV infusion on days 1, 8, and 15 of a 28-day cycle.
  Pelareorep: Pelareorep 4.5 x 10^10 TCID50 1-hour IV infusion days 1, 2, 8, 9, and 15, 16 of a 28-day cycle.
- Pelareorep + Paclitaxel + Avelumab: Patients receive pelareorep + paclitaxel + avelumab.
  Paclitaxel: Paclitaxel 80 mg/m^2 1-hour IV infusion on days 1, 8, and 15 of a 28-day cycle.
  Pelareorep: Pelareorep 4.5 x 10^10 TCID50 1-hour IV infusion days 1, 2, 8, 9, and 15, 16 of a 28-day cycle.
  Avelumab: Avelumab 10 mg/kg (not more than 800 mg) 1-hour IV infusion days 3 and 17 of a 28-day cycle.
Period: Overall Study
Arm/Group | Paclitaxel | Pelareorep + Paclitaxel | Pelareorep + Paclitaxel + Avelumab
Started | 15 | 16 | 17
Completed | 15 | 16 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is an open-label randomized Phase 2, 3-cohort study for patients with hormone receptor (HR)-positive (HR+)/ Human Epidermal Growth Factor Receptor 2 (HER2)-negative (HER2-), endocrine-refractory metastatic breast cancer.
Groups:
- Pelareorep: Patients receive paclitaxel alone.
  Paclitaxel: Paclitaxel 80 mg/m^2 1-hour IV infusion on days 1, 8, and 15 of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Pelareorep | Pelareorep + Paclitaxel | Pelareorep + Paclitaxel + Avelumab | Total
Number analyzed (Participants) | 15 | 16 | 17 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 14 | 14 | 38
  >=65 years | 5 | 2 | 3 | 10
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [46 to 74] | 52.8 [38 to 71] | 55.1 [37 to 70] | 56.2 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 17 | 48
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 14 | 13 | 13 | 40
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 4 | 8
  White | 12 | 12 | 13 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate at week 16 according to RECIST V1.1
Time Frame: at week 16
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Pelareorep | Pelareorep + Paclitaxel | Pelareorep + Paclitaxel + Avelumab
Number analyzed (Participants) | 15 | 16 | 17
percentage of participants | 20 [7.6 to 39.3] | 31.3 [16.1 to 50.4] | 14.3 [3.9 to 33.7]

2. Other Pre Specified Outcome: The Number of Patients With Adverse Events and Serious Adverse Events
Description: Graded by the NCI CTCAE v. 5.0.
Time Frame: From first day of study treatment to 30 days after of last day of study treatment; up to 27 months
Population: The Safety Analysis set comprises all patients who received any amount of study treatment. A total of 48 patients were enrolled. In the Paclitaxel Arm, 15 patients were randomized / 12 patients recieved study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Paclitaxel: Paclitaxel 80 mg/m2 1-3 hour IV infusion weekly days 1, 8, and 15
- Paclitaxel + Pelareorep: Paclitaxel 80 mg/m2 1-3 hour IV infusion weekly days 1, 8, and 15; plus Pelareorep 4.5 x 1010 TCID50 1-hour IV infusion days 1, 2, 8, 9, 15, and 16
- Paclitaxel + Pelareorep + Avelumab: Paclitaxel 80 mg/m2 1- 3 hour IV infusion weekly days 1, 8, and 15; plus Pelareorep 4.5 x 1010 TCID50 1-hour IV infusion days 1, 2, 8, 9, 15, and 16; and Avelumab 10 mg/kg (not more than 800 mg) 1-hour IV infusion days 3 and 17
Arm/Group | Paclitaxel | Paclitaxel + Pelareorep | Paclitaxel + Pelareorep + Avelumab
Number analyzed (Participants) | 12 | 16 | 17
Participants | 12 | 16 | 17

3. Other Pre Specified Outcome: Changes in the Peripheral and Tumor T Cell Clonality.
Description: Assessed by T cell receptor (CDR3 variable chain) sequencing in all patients.
Time Frame: Up to 2 years of study treatment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Response Rate
Description: Overall response rate according to RECIST V1.1
Time Frame: Up to 2 years of study participation
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Overall Survival
Description: Overall Survival assessed at end of study
Time Frame: Up to 2 years of study participation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 27 months
Arm/Group | Pelareorep | Pelareorep + Paclitaxel | Pelareorep + Paclitaxel + Avelumab
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/12 | 4/16 | 13/17
Other Adverse Events (participants affected / at risk) | 12/12 | 16/16 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pelareorep (N=12) | Pelareorep + Paclitaxel (N=16) | Pelareorep + Paclitaxel + Avelumab (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pelareorep (N=12) | Pelareorep + Paclitaxel (N=16) | Pelareorep + Paclitaxel + Avelumab (N=17)
Fatigue (General disorders) | 5 (5) | 12 (12) | 8 (8)
Pyrexia (General disorders) | 1 (1) | 9 (9) | 13 (13)
Chills (General disorders) | 0 (0) | 7 (7) | 6 (6)
Oedema peripheral (General disorders) | 2 (2) | 6 (6) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 4 (4) | 5 (5)
Pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 2 (2) | 7 (7) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 7 (7) | 9 (9)
Neutrophil count decreased (Investigations) | 3 (3) | 5 (5) | 11 (11)
White blood cell count decreased (Investigations) | 3 (3) | 3 (3) | 11 (11)
Alanine aminotransferase increased (Investigations) | 4 (4) | 6 (6) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 4 (4) | 3 (3)
Lymphocyte count decreased (Investigations) | 3 (3) | 3 (3) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 6 (6)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 2 (2)
Blood creatine increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 8 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (9) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 6 (6) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 9 (9)
Proteinuria (Renal and urinary disorders) | 2 (2) | 7 (7) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04215146/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT04215146/SAP_001.pdf